CLINICAL TRIAL: NCT02956993
Title: A Phase 1, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Study of Vonapanitase Administered Following Angioplasty of a Distal Popliteal, Tibial or Peroneal Artery in Patients With Peripheral Artery Disease
Brief Title: Safety/Feasibility of Vonapanitase Following Angioplasty for Patients With Peripheral Artery Disease (PAD) Below the Knee (BTK)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Proteon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRT-201-115
Record Dates: First submitted 2016-11-03; First posted 2016-11-07 (Estimated); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Peripheral Artery Disease
Keywords: peripheral artery disease; PAD; vonapanitase; critical limb ischemia; CLI; tibial artery; stenosis; distal popliteal artery; peroneal artery; below the knee; BTK; elastase; chymotrypsin-like elastase 1; CELA1; PRT-201
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia; Constriction, Pathologic | interventions — cholesterol-binding protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vonapanitase (Active Comparator): Vonapanitase administered to the distal popliteal, tibial or peroneal artery using a micro-infusion catheter.
  Interventions: Drug: vonapanitase
- Placebo (Placebo Comparator): Placebo administered to the distal popliteal, tibial or peroneal artery using a micro-infusion catheter.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: vonapanitase
  Other Names: PRT-201
  Arms: Vonapanitase
Drug: Placebo
  Arms: Placebo

SUMMARY:
The research study is designed to assess the technical feasibility and safety of a perivascular injection of vonapanitase delivered via micro-infusion catheter to the distal popliteal, tibial or peroneal arteries immediately following successful angioplasty.

ELIGIBILITY:
Screening: Initial study inclusion criteria

1. Age of at least 18 years.
2. Clinical diagnosis of PAD secondary to atherosclerosis affecting a lower limb.
3. Rutherford category 3-5.
4. De novo lesion, not previously treated by angioplasty, atherectomy or stenting.
5. Scheduled to undergo angioplasty of the distal popliteal, tibial or peroneal arteries.
6. If female and of childbearing potential (premenopausal and not surgically sterile) must have a negative pregnancy test at the screening visit and be willing to use contraception from the time of the screening visit to 1 week following study drug administration. Acceptable methods of birth control include abstinence, barrier methods with spermicide, implants, injectables, oral contraceptives, intra-uterine device, or a vasectomized partner.
7. Ability to understand and comply with the requirements of the entire study and communicate with the study team.
8. Ability to provide written informed consent using a document that has been approved by the required institutional review board.

   Procedure: Study inclusion criteria to be determined at the time of the angioplasty procedure
9. Atherosclerotic lesion with >50% stenosis in the popliteal (distal to the center of the knee joint space, the P3 segment), tibial or peroneal artery prior to angioplasty.
10. Successful revascularization without the use of stenting of the target lesion; no flow limiting dissection and <30% residual lumen stenosis as compared with an adjacent non-diseased lumen diameter.

Exclusion Criteria Screening: Initial study exclusion criteria

1. Patients in whom arterial insufficiency in the lower extremity is the result of an immunologic or inflammatory non-atherosclerotic disorder (e.g., Buerger's disease, vasculitis).
2. Planned above ankle amputation on ipsilateral limb within 4 weeks of study drug administration.
3. Prior or planned stenting of the target lesion.
4. Deep vein thrombosis within the past 3 months.
5. Known bleeding disorder.
6. Known hypercoagulable state (e.g., protein C deficiency, factor V Leiden, prothrombin G20210A mutation).
7. Platelet count <130K, hematocrit <30%, bilirubin or ALT >3.0 times the upper limit of normal.
8. Renal failure with existing dependence on dialysis or an eGFR by MDRD calculation of < 20 mL/min/1.73 m2.
9. Pregnancy, lactation or plans to become pregnant during the course of the study.
10. Presence of any significant medical condition that might significantly confound the collection of safety and efficacy data in this study.
11. Malignancy or treatment for malignancy within the previous 12 months with the exception of localized basal cell or squamous cell skin cancer, or any cancer in situ.
12. Treatment with any investigational drug within the previous 30 days or investigational antibody therapy within 90 days prior to signing informed consent.
13. Known allergy to radiocontrast agents.

    Procedure:

    Exclusion criteria to be determined at the time of the angioplasty procedure
14. Reference vessel diameter < 2 mm and > 8 mm.
15. Severe concentric medial calcification of the target lesion thought to interfere with study drug delivery to the adventitia based on fluoroscopic appearance.
16. Aneurysm in the target vessel.
17. Failure to cross the target lesion with a guide wire; however subintimal wire crossing is allowed.
18. Stenting of the target lesion.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-11; Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 6 months following study drug administration
  Safety assessments include physical exams and routine serum chemistry and hematology tests
Technical success of perivascular injection | Intraprocedural
  Technical success of study drug administration will be assessed by the extent of circumferential and longitudinal coverage of the artery using a protocol-defined assessment scale

OTHER OUTCOMES:
Minimum lumen diameter [MLD] | Intraprocedural and 6 months following study drug administration
Minimum lumen area [MLA] | Intraprocedural and 6 months following study drug administration
Incidence of arterial occlusion | 14 days and 6 months following study drug administration
Rutherford category | 14 and 28 days, and 6 months following study drug administration
Ankle-brachial index [ABI] | 14 days and 6 months following study drug administration
Vascular Quality of Life Questionnaire-6 [VascuQol-6 | 14 days and 6 months following study drug administration

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - VA Medical Center Long Beach, Long Beach, California
  - VA Eastern Colorado Healthcare System, Denver, Colorado
  - UF Health at the University of Florida, Gainesville, Florida
  - Boston Medical Center, Boston, Massachusetts
  - Steward St. Elizabeth's Medical, Boston, Massachusetts
  - Metro Health Hospital, Wyoming, Michigan
  - Cardiothoracic and Vascular Surgeons, Austin, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin